CLINICAL TRIAL: NCT05201612
Title: Phase II Trial of Pembrolizumab and Olaparib in Homologous-recombination Deficient (HRD) Advanced Colorectal Cancer (CRC).
Brief Title: Pembrolizumab and Olaparib in Homologous-recombination Deficient (HRD) Advanced Colorectal Cancer (CRC).
Acronym: PEMBROLA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Collaborators: Merk Sharp & Dohme España S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-2102; 2021-003767-10 (EudraCT Number)
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: HRD deficient colorectal cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — olaparib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: All patients will receive pembrolizumab 200 mg IV every 3 weeks and olaparib 300 mg, po, bid continuously until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab plus olaparib (Experimental): Treatment cycles will be 21 days in length. All participants will receive treatment as follows:
  Olaparib 300 mg, orally (po), twice a day (BID) continuously. Pembrolizumab 200 mg, intravenously (IV), every 21 days. Treatment will be continued in the absence of disease progression, unacceptable toxicity, withdrawal of consent or death. Pembrolizumab will be administered up to a maximum of 2 years (35 cycles).
  Interventions: Drug: Olaparib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Olaparib — Olaparib 300 mg, orally (po), twice a day (BID) continuously
  Other Names: Lynparza
Drug: Pembrolizumab — Pembrolizumab 200 mg, intravenously (IV), every 21 days. Max 2 years (i.e. 35 cycles)
  Other Names: Keytruda

SUMMARY:
Colorectal Cancer (CRC) is a leading cause of cancer-related death. Around 30% of patients present with advanced disease and 50% of those that attempt curative surgery will eventually relapse. The potential synergism of combining PARP inhibitor and PD-L1 is based on the hypothesis that pharmacological inhibition of PARP by olaparib will result in enhanced immunogenicity which can be further enhanced with an immune checkpoint inhibitor such as pembrolizumab. This may occur through a number of mechanisms, such as increased production of cytokines and chemokines that have the potential to promote antitumour immunity, upregulation of surface receptors which render tumour cells more visible to detection by cytotoxic T cells thereby leading to death of tumour cells and release of neoantigens, that help promote antigen presentation and immune priming. This hypothesis is supported by preclinical studies in mouse models of cancer, demonstrating that administration of a PARP inhibitor to sensitive tumour types resulted in increased T cell infiltration and immune activation within tumours.

The primary hypothesis is that Olaparib and pembrolizumab combination will lead to an increase in objective response rate in patients with refractory metastatic colorectal cancer (mCRC) with DNA homologous-recombination-repair deficiency (HRD) from 1.5% in benchmark studies to up to >10%. The primary objective of the study is to determine the objective response rate (ORR) of pembrolizumab in combination with olaparib, assessed by the investigator per RECIST criteria version 1.1. Secondary objectives include efficacy in terms of disease control rate (DCR), progression-free survival (PFS), overall survival (OS) and duration of response (DOR); safety and an exploratory study of biomarkers associated with treatment efficacy and disease prognosis.

DETAILED DESCRIPTION:
This study is a phase 2, open-label, multicentric, single arm trial designed to evaluate the response to olaparib in combination with pembrolizumab in patients with metastatic colorectal cancer (mCRC) with homologous-recombination repair deficiency (HRD), defined as the presence of a BRCA deleterious mutation and/or a low RAD51 score (cut-off <10% ) [Castroviejo-Bermejo, 2018].

Patients will be required to provide a sample of the most recent archival tumor tissue for HRD determination. A functional score evaluating HRD deficiency will be performed, the RAD51 score. This score will be determined in FFPE tumor samples. Oxaliplatin-sensitivity and a low RAD51 score (cut-off <10%) will be required for patients to continue the screening process.

Oxaliplatin-sensitivity is defined as a progression free survival ≥ 9 months in the first line setting, having received at least 8 cycles of FOLFOX (fluorouracil, folinic acid and oxaliplatin) or 6 cycles of XELOX (capecitabine and oxaliplatin) treatment as first line therapy.

All patients will undergo screening assessments within 4 weeks prior to enrollment. Screening assessments will include demographics and medical history, prior anticancer treatments and sensibility to oxaliplatin therapy, prior and current medications, 12-lead ECG, ECOG performance status, hematology and serum/plasma chemistry, urinalysis, physical examination, vital signs measurements, and baseline radiologic assessment by whole body computed tomography (CT).

All patients included in the study will undergo the Myriad MyChoice HRD test, but no specific cut-off value will be requested to participate in the trial.

Treatment cycles will be 21 days in length. All participants will receive treatment as follows:

Olaparib 300 mg, orally (po), twice a day (BID) continuously. Pembrolizumab 200 mg, intravenously (IV), every 21 days. Treatment will be continued in the absence of disease progression, unacceptable toxicity, withdrawal of consent or death. Pembrolizumab will be administered up to a maximum of 2 years (35 cycles).

All patients will be monitored for efficacy as well as safety throughout this phase. Assessments will include physical examination, vital signs and weight assessment, hematology, serum chemistry, urinalysis, concomitant medications, ECOG performance status, disease status assessment, 12-lead ECG, AEs with any associated therapies and procedures, study drug administration and accountability.

Disease response to study treatment will be evaluated by imaging methods, with tumor scans being done every 9 weeks of treatment (± 7 days). Disease progression will be determined by RECIST v1.1. Patients experiencing disease progression by RECIST v1.1, as assessed by the investigator, will be discontinued from study treatment and continue follow-up. However, if the patient has met criteria for radiologic progression by RECIST, but is still benefiting from the study drugs, according to the investigator, the decision to continue will be made jointly between the investigator and the sponsor.

Upon treatment discontinuation (with the exception of withdrawal of consent or death), patients will have an End of Treatment Visit. All patients will be followed for at least 28 days after the last dose of study drug and will then be followed every 3 months for survival.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants must be at least 18 years of age on the day of signing informed consent and have a histologically confirmed diagnosis of colorectal cancer.
2. Have an unresectable locally-advanced or metastatic colorectal cancer and have progressive disease confirmed by radiologic assessment.
3. Have provided an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
4. Have DNA HRD defined as either having a BRCA known deleterious mutation (somatic or germinal) and/or RAD 51 score < 10%.
5. Have received at least 2 and no more than 4 prior lines of systemic therapy (including adjuvant treatment). Patients must have received at least: fluoropyrimidines, oxaliplatin and irinotecan, with or without anti-VEGF or anti-EGFR therapy if RAS wild type.
6. Must be oxaliplatin-sensitive defined as having received a minimum of 8 cycles of FOLFOX (fluorouracil, folinic acid and oxaliplatin) or 6 cycles of XELOX (capecitabine and oxaliplatin) as first line therapy, and a progression free survival ≥ 9 months in the first line setting.
7. Patients with both MSS or MSI-H advanced colorectal cancer will be suitable to participate in the trial.
8. The participant (or legally acceptable representative if applicable) provides written informed consent to participate in the trial.
9. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions after radiotherapy.
10. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
11. Have adequate organ function. Blood samples must be collected within 7 days prior to the start of study intervention.
12. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 28 days prior to any study treatment administration plus an additional 180 days after the last dose of study treatment and refrain from donating sperm during this period.
13. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
    2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 180 days after the last dose of study treatment.

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137) or with any PARP inhibitor.
2. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

   * Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
   * Participation in an observational (non-interventional) study is allowed.
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.

   * Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible
   * If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   -In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
6. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
9. Has known CNS metastases and/or carcinomatous meningitis.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab or olaparib and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease of any etiology.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV) infection. No HIV testing is required
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.

    No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
17. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
18. Current, clinically relevant bowel obstruction, including sub-occlusive disease, related to underlying disease or any other non-reversible cause.
19. Patient has any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of trial treatment.
22. Has had an allogenic tissue/solid organ transplant.
23. Other severe acute or chronic medical condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Throughout the study period, approximately 10 months per patient from first study dose.
  Objective response rate (ORR) according to investigator assessment following RECIST criteria version 1.1. ORR has been defined as the number of participants with a best overall response (BOR) of confirmed CR or PR divided by the number of enrolled participants. BOR is defined as the best response designation, determined by the investigator, recorded between the date of treatment start and the date of objectively documented progression per RECIST 1.1 or, the date of initiation of subsequent anti-cancer therapy, whichever occurs first. Complete or partial responses may be claimed only if the criteria for each are met at a subsequent time point of ≥ 4 weeks later.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Throughout the study period, approximately 10 months per patient from first study dose.
  DCR is defined as the number of participants with a best overall response of confirmed stable disease, CR or PR divided by the number of enrolled participants. Best overall response will be determined by investigator, recorded between the date of treatment start and the date of objectively documented progression per RECIST 1.1 or, the date of initiation of subsequent anti-cancer therapy, whichever occurs first.
Progression-free survival (PFS) | Throughout the study period, approximately 10 months per patient from first study dose.
  PFS is defined as the time from the allocation date to the date of the first documented tumor progression per RECIST 1.1, or death due to any cause. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments will be censored on the beginning of treatment date. Median values will be provided
Overall survival (OS) | Throughout the study period, approximately 10 months per patient from first study dose.
  OS is defined as the time from treatment allocation to the date of death due to any cause. OS with 95% CIs will be estimated using Kaplan-Meier methodology. Median values will be provided.
Duration of response (DOR) | Throughout the study period, approximately 10 months per patient from first study dose.
  DOR will be defined as the time from the date of first documented response (CR/PR) as per RECIST 1.1 as assessed by the investigator until the date of documented progression or death in the absence of disease progression, the end of response will coincide with the date of progression or death from any cause. The time of the initial response will be defined as the latest of the dates contributing towards the first visit response of PR or CR. Median values will be provided.

OTHER OUTCOMES:
HRD score as per the Myriad MyChoice HRD test | Throughout the study period, approximately 10 months per patient from first study dose.
  Percentage of HRD positive patients and median HRD score among responders and non responders (patients stratified according to ORR)
Biomarker molecular substudy | Throughout the study period, approximately 10 months per patient from first study dose.
  Percentage of patients presenting molecular alterations of prognostic value (i.e. BRCA deleterious mutations or HRD deficiency among others)

CONTACTS AND LOCATIONS:
Overall Officials: Rocío García Carbonero, M.D.; Ph.D., Principal Investigator — Hospital Universitario 12 de Octubre; María del Carmen Riesco Martinez, M.D.; Ph.D., Principal Investigator — Hospital Universitario 12 de Octubre
Locations (15):
- Spain (15):
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida, Catalonia
  - Hospital de Sabadell, Sabadell, Catalonia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital General Universitario de Elche, Elche, Valencia
  - Fundacion Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia